CLINICAL TRIAL: NCT03416530
Title: ONC201 in Newly Diagnosed Diffuse Intrinsic Pontine Glioma and Recurrent/Refractory Pediatric H3 K27M Gliomas
Brief Title: ONC201 in Pediatric H3 K27M Gliomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor terminated the study to prioritize enrollment in a randomized Phase 3 trial of ONC201 in an earlier setting. This decision was unrelated to any safety concerns with dordaviprone (ONC201).
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Oncoceutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC014
Record Dates: First submitted 2018-01-23; First posted 2018-01-31 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Glioma, Malignant
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioma | interventions — TIC10 compound

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- A (recurrent/refractory H3 K27M-mutant glioma) (Experimental): Pediatric patients with relapsed/refractory glioma who are positive for the H3 K27M mutation (positive testing in CLIA laboratory) and have completed at least one line of prior therapy. Evidence of progression is not required so that ONC201 may be administered to patients in the maintenance setting or to patients with recurrent/refractory disease.
  Interventions: Drug: Dordaviprone (ONC201)
- B (newly diagnosed DIPG) (Experimental): Pediatric patients with newly diagnosed diffuse intrinsic pontine glioma (DIPG), defined as tumors with a pontine epicenter and diffuse involvement of the pons, are eligible with or without histologic confirmation. If H3 K27M status of tumor is unknown or archival tumor tissue is not available, then patients must agree to submit a post-mortem biopsy specimen.
  Interventions: Drug: Dordaviprone (ONC201)
- C (midline glioma) (Experimental): Pediatric patients with midline gliomas are eligible with or without histologic confirmation and must be eligible for tumor biopsy as deemed by the site Investigator.
  Interventions: Drug: Dordaviprone (ONC201)
- D (recurrent H3 K27M-mutant glioma; CSF obtained) (Experimental): Pediatric patients with recurrent glioma who are positive for the H3 K27M mutation (positive testing in CLIA laboratory), have completed at least one line of prior therapy, must be willing to undergo serial lumbar puncture to obtain cerebrospinal fluid (CSF), and must be scheduled to undergo sedated MRIs.
  Interventions: Drug: Dordaviprone (ONC201)
- E (H3 K27M-mutant glioma or DIPG; liquid formulation) (Experimental): Patients with glioma who are positive for the H3 K27M mutation (positive testing in CLIA laboratory) or have diagnosed diffuse intrinsic pontine glioma (DIPG), defined as tumors with a pontine epicenter and diffuse involvement of the pons, are eligible with or without histologic confirmation. Patients must be 2-12 weeks from completion of first-line radiation. Patients administered liquid formulation of dordaviprone (ONC201) in Ora-Sweet.
  Interventions: Drug: Dordaviprone (ONC201)
- F (recurrent/refractory, progressive high-grade H3 K27M-mutant glioma) (Experimental): Pediatric patients with relapsed/refractory, histologically confirmed high-grade glioma with a known H3 K27M mutation, evidence of progressive disease contrast-enhanced brain MRI as defined by RANO-HGG criteria. Prior therapy with at least radiotherapy is required.
  Interventions: Drug: Dordaviprone (ONC201)
- G (recurrent/refractory H3 K27M-mutant glioma; dosing twice weekly) (Experimental): Pediatric patients with glioma who are positive for the H3 K27M mutation (positive testing in CLIA laboratory) and have completed at least one line of prior therapy will be enrolled to define the RP2D for single agent dordaviprone (ONC201) given on two consecutive days of each week.
  Interventions: Drug: Dordaviprone (ONC201)

INTERVENTIONS:
Drug: Dordaviprone (ONC201) — Dordaviprone is a brain-penetrant, small-molecule imipridone that acts as a mitochondrial caseinolytic protease P (ClpP) agonist and a dopamine receptor D2 (DRD2) antagonist.

SUMMARY:
This was a Phase 1, open label, multicenter, 8-arm, dose escalation study of dordaviprone (ONC201) in pediatric patients with newly diagnosed diffuse intrinsic pontine glioma (DIPG) and recurrent/refractory H3 K27M-mutant gliomas.

The primary endpoint of this study was to determine the recommended Phase 2 dose (RP2D) of dordaviprone (ONC201) in pediatric glioma patients as a single agent in combination with radiation.

DETAILED DESCRIPTION:
This study was to include 8 arms; the intention for each arm is summarized below:

* Arm A: To define the RP2D for single agent dordaviprone (ONC201) in pediatric patients with glioma who are positive for the H3 K27M mutation and have completed at least 1 line of prior therapy.
* Arm B: To define the RP2D for dordaviprone (ONC201) in combination with radiation in pediatric patients with newly diagnosed DIPG.
* Arm C: To determine intratumoral drug concentrations and biomarker expression in pediatric patients with midline gliomas.
* Arm D: To determine H3 K27M DNA levels and drug concentrations in the cerebral spinal fluid (CSF) of pediatric patients with H3 K27M-mutant glioma.
* Arm E: To define the RP2D for single agent dordaviprone (ONC201) when administered as a liquid formulation in Ora-Sweet to pediatric patients with DIPG and/or H3 K27M-mutant glioma.
* Arm F: A dose expansion cohort to confirm the safety and estimate the efficacy of dordaviprone (ONC201) in recurrent H3 K27M-mutant glioma at the RP2D.
* Arm G: To define the RP2D for single agent dordaviprone (ONC201) when administered on 2 consecutive days of each week in pediatric patients with H3 K27M-mutant glioma who have completed at least 1 line of prior therapy.
* Arm H: To assess intra-tumoral concentrations following twice weekly dosing of dordaviprone (ONC201) in 2 cohorts: pediatric patients with DIPG and pediatric patients with thalamic gliomas. *Note: This arm did not enroll any patients.

Pediatric patients in Arms A through F received dordaviprone (ONC201) once weekly. Patients in Arms C, D, E, and F received dordaviprone (ONC201) at the RP2D determined in either Arm A or Arm B. Pediatric patients in Arm G received dordaviprone (ONC201) twice weekly on 2 consecutive days.

Safety was also assessed, with evaluations including the reporting of adverse events, as well as measurements of vital signs, electrocardiograms, and clinical laboratory results.

This study was terminated by an administrative protocol amendment (17 January 2023). The decision to terminate the study was not related to any safety concerns with dordaviprone (ONC201). Before the study was terminated a total of 134 patients were enrolled and had received at least 1 dose of dordaviprone (ONC201). At the time of the administrative protocol amendment, patient enrollment was completed in Arms A, B, C, D, E, and G, and patient enrollment was stopped prior to reaching the targeted enrollment in Arms F and H.

ELIGIBILITY:
Inclusion Criteria:

1. 2 to less than 19 years of age.
2. Patient body weight must be above the minimum necessary for the patient to receive the ONC201 dose indicated for the currently enrolling dose level. The minimum body weight ranges from 10-27.5kg depending on the dose level.
3. Arm A and G: Patients with glioma who are positive for the H3 K27M mutation (positive testing in CLIA laboratory) and have completed at least one line of prior therapy. Evidence of progression is not required so that ONC201 may be administered to patients in the maintenance setting or to patients with recurrent disease. No more than two episodes of recurrence from radiotherapy and/or chemotherapy are allowed. Use of bevacizumab solely for treatment of radiation necrosis, pseudoprogression, or treatment effect will not be considered a recurrence. Post-mortem biopsy is required if H3 K27M status of tumor is unknown and archival tumor tissue not available.

   Arm B: Patients with newly diagnosed diffuse intrinsic pontine glioma (DIPG), defined as tumors with a pontine epicenter and diffuse involvement of the pons, are eligible with or without histologic confirmation. Post-mortem biopsy is required if H3 K27M status of tumor is unknown and archival tumor tissue not available.

   Arm C: Patients with midline gliomas are eligible with or without histologic confirmation and must be eligible for tumor biopsy as deemed by the site Investigator.

   Arm D: Patients with recurrent glioma who are positive for the H3 K27M mutation (positive testing in CLIA laboratory), have completed at least one line of prior therapy, must be willing to undergo serial lumbar puncture to obtain cerebrospinal fluid (CSF), and must be scheduled to undergo sedated MRIs. Local anesthesia for spinal tap is also allowed. Evidence of progression is not required so that ONC201 may be administered to patients in the maintenance setting or to patients with recurrent disease. No more than two prior episodes of recurrence from radiotherapy and/or chemotherapy are allowed. Use of bevacizumab solely for treatment of radiation necrosis, pseudoprogression, or treatment effect will not be considered a recurrence. Spinal tap should not be performed if treating clinician or lumbar puncture proceduralist has concern of signs of elevated intracranial pressure, including recent worsening in headache or somnolence.

   Arm E: Patients with glioma who are positive for the H3 K27M mutation (positive testing in CLIA laboratory) or have diagnosed diffuse intrinsic pontine glioma (DIPG), defined as tumors with a pontine epicenter and diffuse involvement of the pons, are eligible with or without histologic confirmation. Patients must be 2-12 weeks from completion of first-line radiation. Evidence of progression is not required so that ONC201 may be administered to patients in the maintenance setting or to patients with recurrent disease.

   Arm F:

   Pediatric patients with histologically confirmed diagnosis of high-grade glioma in any tumor sample with a known histone H3 K27M mutation identified by IHC or DNA sequencing test performed in a CLIA setting. Evidence of progressive disease on contrast-enhanced brain MRI as defined by RANO-HGG criteria is required. Patients must have had previous therapy with at least radiotherapy.
4. Karnofsky ≥ 50 for patients ≥ 16 years of age, and Lansky ≥ 50 for patients < 16 years of age. For Arm F, Karnofsky ≥ 60 for patients ≥ 16 years of age, and Lansky ≥ 60 for patients < 16 years of age
5. From the projected start of scheduled study treatment, the following time periods must have elapsed: 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies, or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies. For patients who have received radiotherapy, patients in any arm must be at least 2 weeks from the completion of local palliative radiotherapy (re-irradiation for progressive disease or upfront radiation at initial diagnosis). For Arm F, patients must be at least 90 days from prior radiation to the first dose of ONC201unless the progressive lesion is outside of the high-dose radiation target volume or there is unequivocal evidence of progressive tumor on a biopsy specimen.
6. Adequate organ function defined as:

   Bone Marrow:
   * Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3 and
   * Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).

   Renal Function:

   • Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70mL/min/1.73 m2 or normal serum creatinine based on age as shown below or GFR > 70ml/min/1.73m^2: Age < 5 years: 0.8 mg/dL maximum Age 5 to < 10 years: 1.0 mg/dL maximum Age 10 to < 15 years: 1.2 mg/dL maximum Age > 15 years: 1.5 mg/dL maximum

   Liver Function:
   * Total Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of institutional normal and
   * SGPT (ALT) ≤ 110 U/L and
   * Serum albumin ≥ 2 g/dL.

   Neurologic Function:

   • Patients with seizure disorder may be enrolled if seizure disorder is well controlled.
7. Ability to understand a written informed consent document, and the willingness to sign it. Assent will be obtained when appropriate based on the subjects age.
8. All adverse events Grade > 1 related to prior therapies (chemotherapy, radiotherapy, and/or surgery) must be resolved to grade 1 or baseline, except for alopecia and sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment, are acceptable.
9. For patients post pubertal: Female patients must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. Male patients must be surgically sterile or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. The decision of effective contraception will be based on the judgment of the principal investigator.
10. Corticosteroid dose must be stable or decreasing for at least 3 days prior to the baseline CT or MRI scan.
11. MRI brain and entire spine MRI within 14 days prior to start of study drug for Arms A, B, C, E, F and G. Subjects undergoing screening for Arm D must have an MRI of brain and entire spine within 3 months prior to start of study drug. Subjects in Arm D will have a baseline MRI of brain and spine with lumbar puncture after study consent is signed and other eligibility criteria are fulfilled.
12. For Arms A, B, C, D, F and G: Ability to swallow and retain orally administered capsules.
13. Archival tumor specimen: Subjects in all arms must submit at least 5 unstained slides from a tumor specimen that harbors H3 K27M mutation if archival tissue is available. For subjects in Arms A, B, E or G, if no archival tumor tissue is available, or if H3 K27M status of tumor is unknown, then subjects must agree to submit a post-mortem biopsy specimen. Subjects in Arm C do not require prior tumor biopsy or confirmation of the presence of the H3 K27M mutation. Subjects in Arm D must have confirmation of the presence of the H3 K27M mutation in any glioma sample prior to enrollment. Subjects in Arm F must submit at least 5 unstained slides from a tumor specimen that harbors H3 K27M mutation. Note that the H3 K27M mutation is often reported as H3 K28M in gene sequencing assays.

Exclusion Criteria:

1. For Arms A, B, D, E, F and G: Evidence of diffuse leptomeningeal disease or evidence of CSF dissemination.
2. Current or planned participation in a study of another investigational agent or using an investigational device.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ONC201 or its excipients.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
5. Any known clinically significant active infection including bacterial, fungal or viral including hepatitis B (HBV), hepatitis C (HCV) or any underlying disease or in the recent past which could compromise enrollment and safety of the patient
6. Known history of cardiac arrhythmias including atrial fibrillation, tachyarrhythmias or bradycardia, unless arrhythmia is controlled and after Cardiology has cleared patient to receive ONC201. Receiving therapeutic agents known to prolong QT interval will be excluded, however the use of Zofran is permitted. History of CHF, or MI or stroke in the last 3 months will be excluded.
7. Active illicit drug use or diagnosis of alcoholism.
8. Known additional malignancy that is progressing or requires active treatment within 3 years of start of study drug.
9. Concomitant use of potent CYP3A4/5 inhibitors during the treatment phase of the study and within 72 hours prior to starting study drug administration.
10. Concomitant use of potent CYP3A4/5 inducers, which include enzyme inducing antiepileptic drugs (EIAEDs) (see Appendix B), during the treatment phase of the study and within 2 weeks prior to starting treatment. Concurrent dexamethasone is allowed.
11. For Arm F: Exclusively non-contrast-enhancing disease or primary malignant lesion located in the pons or spinal cord.
12. For Arm F: Atypical non-astrocytic histologies such as ependymoma, ganglioma and pleomorphic xanthoastrocytoma, pilocytic astrocytoma, or pilocytic astrocytoma and subependymal giant cell astrocytoma (SEGA).
13. Prior treatment with ONC201

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
RP2D | 28 days
  Determination of recommended Phase 2 dose (RP2D) as a single agent or in combination with radiation

CONTACTS AND LOCATIONS:
Overall Officials: Allen Mellemed, MD, Study Director — Chimerix, Inc.
Locations (8):
- United States (8):
  - UCSF, Benioff Children's Hospital, San Francisco, California
  - Miami Cancer Institute, Miami, Florida
  - Children's Healthcare of Atlanta, Emory University School of Medicine, Atlanta, Georgia
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - New York University, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Arrillaga-Romany I, Gardner SL, Odia Y, Aguilera D, Allen JE, Batchelor T, Butowski N, Chen C, Cloughesy T, Cluster A, de Groot J, Dixit KS, Graber JJ, Haggiagi AM, Harrison RA, Kheradpour A, Kilburn LB, Kurz SC, Lu G, MacDonald TJ, Mehta M, Melemed AS, Nghiemphu PL, Ramage SC, Shonka N, Sumrall A, Tarapore RS, Taylor L, Umemura Y, Wen PY. ONC201 (Dordaviprone) in Recurrent H3 K27M-Mutant Diffuse Midline Glioma. J Clin Oncol. 2024 May 1;42(13):1542-1552. doi: 10.1200/JCO.23.01134. Epub 2024 Feb 9. PMID 38335473
- [Derived] Cantor E, Wierzbicki K, Tarapore RS, Ravi K, Thomas C, Cartaxo R, Nand Yadav V, Ravindran R, Bruzek AK, Wadden J, John V, May Babila C, Cummings JR, Rahman Kawakibi A, Ji S, Ramos J, Paul A, Walling D, Leonard M, Robertson P, Franson A, Mody R, Garton HJL, Venneti S, Odia Y, Kline C, Vitanza NA, Khatua S, Mueller S, Allen JE, Gardner SL, Koschmann C. Serial H3K27M cell-free tumor DNA (cf-tDNA) tracking predicts ONC201 treatment response and progression in diffuse midline glioma. Neuro Oncol. 2022 Aug 1;24(8):1366-1374. doi: 10.1093/neuonc/noac030. PMID 35137228